CLINICAL TRIAL: NCT06953960
Title: A Phase 1/2, Open-Label, Platform Study to Evaluate Safety and Efficacy of the BCL-2 Inhibitor Surzetoclax (ABBV-453) Given as Monotherapy or in Combination With Antimyeloma Regimens in Subjects With Multiple Myeloma
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Oral ABBV-453 Alone or in Combination With Subcutaneous and/or Oral Antimyeloma Agents in Adult Participants With Multiple Myeloma (MM)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-275; 2024-517140-65 (Other: EU CT)
Record Dates: First submitted 2025-04-17; First posted 2025-05-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; ABBV-453; Daratumumab; Dexamethasone; Pomalidomide; Cancer
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — daratumumab; Dexamethasone; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Substudy 1: Dose Escalation ABBV-453 Combination (Experimental): Participants will receive various doses of ABBV-453 in combination with daratumumab + dexamethasone, to determine the best dose of ABBV-453, as part of the total 4.5 year study duration.
  Interventions: Drug: ABBV-453; Drug: Daratumumab; Drug: Dexamethasone
- Substudy 1: Dose Expansion and Selection ABBV-453 Combination (Experimental): Participants will receive 1 of 2 doses of ABBV-453 in combination with daratumumab + dexamethasone, as part of the total 4.5 year study duration.
  Interventions: Drug: ABBV-453; Drug: Daratumumab; Drug: Dexamethasone
- Substudy 1: Dose Expansion and Selection Control (Active Comparator): Participants will receive daratumumab, dexamethasone, and pomalidomide, as part of the total 4.5 year study duration.
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Pomalidomide
- Substudy 2: Dose Escalation ABBV-453 Monotherapy (Experimental): Japanese participants will receive various doses of ABBV-453 as a monotherapy, to determine the best dose of ABBV-453, as part of the total 4.5 year study duration.
  Interventions: Drug: ABBV-453

INTERVENTIONS:
Drug: ABBV-453 — Oral Tablet
  Arms: Substudy 1: Dose Escalation ABBV-453 Combination; Substudy 1: Dose Expansion and Selection ABBV-453 Combination; Substudy 2: Dose Escalation ABBV-453 Monotherapy
Drug: Daratumumab — Subcutaneous (SC) Injection
  Arms: Substudy 1: Dose Escalation ABBV-453 Combination; Substudy 1: Dose Expansion and Selection ABBV-453 Combination; Substudy 1: Dose Expansion and Selection Control
Drug: Dexamethasone — Oral Tablet
  Arms: Substudy 1: Dose Escalation ABBV-453 Combination; Substudy 1: Dose Expansion and Selection ABBV-453 Combination; Substudy 1: Dose Expansion and Selection Control
Drug: Pomalidomide — Oral Capsule
  Arms: Substudy 1: Dose Expansion and Selection Control

SUMMARY:
Multiple myeloma (MM) is a plasma cell disease characterized by the growth of clonal plasma cells in the bone marrow. The purpose of this study is to assess the safety and change in disease activity of ABBV-453 in adult participants with relapsed/refractory (R/R) MM. Adverse events and change in disease activity will be assessed.

ABBV-453 is an investigational drug being developed for the treatment of R/R MM. In Substudy 1 there will be a dose escalation phase where participants will receive various doses of ABBV-453 in combination with daratumumab + dexamethasone, to determine the best dose of ABBV-453. This will be followed by a dose expansion and selection phase where participants will receive 1 of 2 doses of ABBV-453 in combination with daratumumab + dexamethasone, or daratumumab + dexamethasone + pomalidomide (only during the expansion phase). In Substudy 2, there will be a dose escalation phase where participants will receive various doses of ABBV-453 alone. Approximately 130 adult participants with R/R MM will be enrolled in the study in approximately 40 sites worldwide.

In Substudy 1 escalation phase, participants will receive oral ABBV-453 tablets in combination with subcutaneous (SC) daratumumab injections + oral dexamethasone tablets and in the expansion phase, will receive oral ABBV-453 tablets in combination with SC daratumumab injections + oral dexamethasone tablets or daratumumab injections + oral pomalidomide + oral dexamethasone tablets. In Substudy 2, Japanese participants will receive oral ABBV-453 tablets. The total study duration is approximately 4.5 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution. The effect of the treatment will be frequently checked by medical assessments, blood tests, and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma (MM) based on standard international myeloma working group (IMWG) diagnostic criteria.
* All participants must have measurable disease per central laboratory with at least 1 of the following assessed within 28 days prior to enrollment:

  * Serum M-protein >= 0.5 g/dL (>= 5g/L); OR
  * Urine M-protein >= 200 mg/24 hours; OR
  * For participants without measurable serum and urine M-protein: Serum free light chain (sFLC) ≥ 10 mg/dL (100 mg/L), provided sFLC ratio is abnormal.
* B-cell lymphoma (BCL)-2 inhibitor treatment naïve.
* t(11;14) positive status and/or BCL2 high status.
* Substudy 1 Dose Escalation Cohorts and Substudy 2:

  -- Must be triple class exposed (PI, IMiD and anti-CD38) and have received 3 to 5 lines of prior antimyeloma therapy, and who have no other appropriate treatment options as deemed by the investigator.
* Substudy 1 Dose Expansion Cohorts:

  * Must be double class exposed (PI, IMiD) and have received 1 to 3 lines of prior antimyeloma therapy.

Exclusion Criteria:

* Major surgery within 4 weeks of study treatment or planned during study participation.
* Active infections: no recent infection requiring systemic treatment that was completed <= 7 days before first dose of study treatment and/or uncontrolled systemic infection.
* Recent infection requiring systemic treatment that was completed <= 7 days before first dose of study treatment and/or uncontrolled active systemic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLT)s of ABBV-453 | Up to Approximately 45 Months
  DLT events are defined as specific clinically significant adverse events or abnormal laboratory values assessed as events regardless of attribution to ABBV-453, except those clearly and incontrovertibly associated with underlying disease or extraneous causes.
Number of Participants with Adverse Events (AE)s | Up to Approximately 4.5 Years
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to Approximately 4.5 Years
  ORR is defined as the percentage of participants with a confirmed partial response (PR), very good partial response, complete response (CR) or stringent complete response (sCR) per Investigator review according to International Myeloma Working Group (IMWG) 2016 criteria.
Progression-Free Survival (PFS) | Up to Approximately 4.5 Years
  PFS is defined as time from first study treatment to the earliest documented disease progression according to IMWG 2016 criteria, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Duration of Response (DOR) | Up to Approximately 4.5 Years
  DOR is defined as the time from the date of achieving the first confirmed sCR/CR/VGPR/PR to the date of recurrence disease progression according to IMWG 2016 criteria, as determined by the investigator, or death of any cause, whichever occurs earlier.
Time-to-Progression (TTP) | Up to Approximately 4.5 Years
  TTP will be defined as the number of days from the date of first dose to the date of earliest disease progression.
Time to Next Treatment | Up to Approximately 4.5 Years
  Time to next treatment will be defined as the number of days from the date of first dose to the date of next treatment.
Minimal Residual Disease (MRD) Negativity | Up to Approximately 4.5 Years
  MRD negativity is defined as having less than 1 myeloma cell that may remain in the bone marrow aspirate per 10^5 nucleated cells and rate of MRD negativity will be determined.
Overall Survival (OS) | Up to Approximately 4.5 Years
  OS is defined as time from first study treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (30):
- United States (4):
  - University of Southern California /ID# 272414, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center - New York - York Avenue /ID# 271214, New York, New York
  - University of North Carolina at Chapel Hill /ID# 272454, Chapel Hill, North Carolina
  - Northwest Medical Specialties Tacoma /ID# 272506, Tacoma, Washington
- Australia (4):
  - Liverpool Hospital /ID# 272002, Liverpool, New South Wales
  - Calvary Mater Newcastle /ID# 272498, Waratah, New South Wales
  - St Vincent's Hospital - Melbourne /ID# 271997, Fitzroy, Victoria
  - Epworth Hospital /ID# 272497, Richmond, Victoria
- Belgium (3):
  - UZ Gent /ID# 271432, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 272382, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 271430, Liège
- France (4):
  - CHU de Montpellier - Hopital Saint Eloi /ID# 275570, Montpellier, Herault
  - Centre Hospitalier Universitaire de Poitiers /ID# 275563, Poitiers, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 275562, Nantes, Pays de la Loire Region
  - Hopital Universitaire Necker Enfants Malades /ID# 275571, Paris, Île-de-France Region
- Israel (5):
  - The Chaim Sheba Medical Center /ID# 271251, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 271252, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 271256, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 271253, Jerusalem
  - Rabin Medical Center. /ID# 272073, Petah Tikva
- Japan (5):
  - Nagoya City University Hospital /ID# 271427, Nagoya, Aichi-ken
  - University Hospital Kyoto Prefectural University of Medicine /ID# 271911, Kyoto, Kyoto
  - The University of Osaka Hospital /ID# 271636, Suita-shi, Osaka
  - Japanese Red Cross Medical Center /ID# 272018, Shibuya-ku, Tokyo
  - The Jikei University Hospital /ID# 272091, Tokyo
- Portugal (3):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil /ID# 275873, Lisbon, Lisbon District
  - Unidade Local de Saude de Braga, EPE /ID# 275853, Braga
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE /ID# 275851, Porto
- Sweden (2):
  - Karolinska University Hospital Solna /ID# 271674, Solna, Stockholm County
  - Sodra Alvsborgs sjukhus /ID# 271822, Borås, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-275